CLINICAL TRIAL: NCT00698464
Title: A Phase I, Open-label, Multi-center, Single Dose Study to Evaluate the Pharmacokinetics and Safety of Subcutaneous Pasireotide (SOM230) in Subjects With Varying Degrees of Hepatic Function
Brief Title: Pharmacokinetics and Safety of Single Subcutaneous Pasireotide (SOM230) in Subjects With Varying Degrees of Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CSOM230B2114
Record Dates: First submitted 2008-06-11; First posted 2008-06-17 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-11

CONDITIONS: Hepatic Cirrhosis; Alcoholism
Keywords: Pasireotide; PK profile,; Single dose; Pasireotide subcutaneous injection; Safety; Mild hepatic impaired patients; Moderate hepatic impaired patients; Severe hepatic impaired patients
MeSH Terms: conditions — Liver Cirrhosis; Alcoholism | interventions — pasireotide

ARMS (1):
- Pasireotide (Experimental)
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide — Single subcutaneous injection of 600 µg of Pasireotide.

SUMMARY:
The purpose of this study is to evaluate the effect of varying degrees of hepatic function (Child-Pugh classification) on the pharmacokinetics and safety of pasireotide s.c. in subjects.

ELIGIBILITY:
Inclusion criteria:

Common Inclusion criteria for all subjects:

* Male or female subjects between 18 and 75 years of age, inclusive.
* Vital signs at screening and baseline which are within normal ranges.
* Subjects must have a BMI between 20 kg/m2 and 30 kg/m2.

Inclusion Criteria for cohort 1:

• Generally healthy subjects as determined by past medical history, physical examination, vital signs, electrocardiogram and standard laboratory tests at screening.

Inclusion Criteria for cohort 2-4:

* Subjects with confirmed cirrhosis by at least one of the following criteria:
* Histologically by prior liver biopsy showing cirrhosis.
* Clinically by physical examination, and/or laboratory data, and/or liver imaging, and/or endoscopic findings.

Exclusion criteria:

Common Exclusion criteria for all subjects:

* Donation or loss of 400 mL or more of blood within eight weeks prior to dosing.
* Subjects with additional active malignant disease within the last five years (with the exception of non-melanoma skin cancers that were not metastatic and have been treated curatively).
* Subjects with abnormal clinical laboratory values (except the clinical laboratory values linked to hepatic dysfunction).
* Any surgical or medical condition that may interfere with the conduct of the study, may jeopardize the subject in case of participation in the study or may significantly alter the absorption, distribution, metabolism or excretion of drugs.
* History of immunocompromise, including a positive HIV test result (ELISA and Western blot). A HIV test will not be required; however, previous medical history will be reviewed
* Female subjects who are pregnant (positive pregnancy test at screening or at baseline) or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control.

Exclusion Criteria for cohort 1:

* Clinical evidence of liver disease or liver injury as indicated by abnormal liver function tests.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result (antibody positive subjects will be allowed if non-viremic).

Exclusion Criteria for cohort 2-4:

* Symptoms or history of encephalopathy (Stage III or worse) within three months prior to dosing.
* Clinical evidence of severe ascites. Exclusion criteria

Common Exclusion criteria for all subjects:

* Donation or loss of 400 mL or more of blood within eight weeks prior to dosing.
* Subjects with additional active malignant disease within the last five years (with the exception of non-melanoma skin cancers that were not metastatic and have been treated curatively).
* Subjects with abnormal clinical laboratory values (except the clinical laboratory values linked to hepatic dysfunction).
* Any surgical or medical condition that may interfere with the conduct of the study, may jeopardize the subject in case of participation in the study or may significantly alter the absorption, distribution, metabolism or excretion of drugs.
* History of immunocompromise, including a positive HIV test result (ELISA and Western blot). A HIV test will not be required; however, previous medical history will be reviewed
* Female subjects who are pregnant (positive pregnancy test at screening or at baseline) or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control.

Exclusion Criteria for cohort 1:

* Clinical evidence of liver disease or liver injury as indicated by abnormal liver function tests.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result (antibody positive subjects will be allowed if non-viremic).

Exclusion Criteria for cohort 2-4:

* Symptoms or history of encephalopathy (Stage III or worse) within three months prior to dosing.
* Clinical evidence of severe ascites.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Determination of the pharmacokinetic profile of single dose of pasireotide s.c. injection. | 5 days

SECONDARY OUTCOMES:
Determination of the safety after a single dose of pasireotide s.c. injection | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticlas, Study Director — Novartis Pharmaceuticlas
Locations (4):
- McGuire Research Institute VAMC, Richmond, Virginia, United States
- Universite Catholique de Louvain, Brussels, Belgium
- Novartis Investigative site, Berlin, Germany
- Novartis Investigative Site, George, South Africa

REFERENCES:
- [Result] Horsmans Y, Hu K, Ruffin M, Wang Y, Song D, Bouillaud E, Wang Y, Mazur D, Botha FP, Heuman DM. Effect of hepatic impairment on the pharmacokinetics of pasireotide (SOM230): results from a multicenter phase I study. J Clin Pharmacol. 2012 Apr;52(4):552-8. doi: 10.1177/0091270011400072. Epub 2012 Jan 26. PMID 22282526
- See also: Novartis Clinical Trial Results on CSOM230B2114 — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2920